CLINICAL TRIAL: NCT03722433
Title: The Efficacy of Probiotic Supplementation in the Reduction of Adverse Effects and Dysbiosis of Helicobacter Pylori Eradication Therapy - A Double Blind, Multi-center Randomized, Placebo Controlled Trial
Brief Title: Probiotics in the Reduction of Adverse Effects and Dysbiosis of H. Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201706036MIPA
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-06

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic plus 14-day sequential therapy (Experimental): D1-D56: probiotics 1 pack bid for 56 days D1-D7: (esomeprazole + amoxicillin bid) for 7 days D8-D14: (esomeprazole + clarithromycin + metronidazole bid) for another 7 days
  Interventions: Drug: Vigiis 101-LAB and sequential therapy
- placebo plus 14-day sequential therapy (Placebo Comparator): D1-D56: placebo 1 pack bid for 56 days D1-D7: (esomeprazole + amoxicillin bid) for 7 days D8-D14: (esomeprazole + clarithromycin + metronidazole bid) for another 7 days
  Interventions: Drug: Placebo and sequential therapy

INTERVENTIONS:
Drug: Vigiis 101-LAB and sequential therapy — Vigiis 101-LAB is the probiotic containing Lactobacillus paracasei subsp. Paracasei, which is the isolate from Taiwanese by Prof. Pan. This strain is resistant to gastric acid and bile acid. Therefore, its survival rate in the gastrointestinal tract could be as high as 95%. Previous studies showed that Vigiis 101-LAB can modulate the gut microbiota, with 10% increase in Bifidobacterium species and 20% reduction in Clostridium difficile.
  Arms: probiotic plus 14-day sequential therapy
Drug: Placebo and sequential therapy — Placebo without Vigiis 101-LAB component
  Arms: placebo plus 14-day sequential therapy

SUMMARY:
The investigators aimed to assess the effect of probiotic supplementation with Vigiis 101-LAB during H. pylori eradication therapy with 14-day sequential therapy in the reduction of adverse effects and the restoration of the dysbiosis.

DETAILED DESCRIPTION:
Backgroud: Helicobacter pylori infection has been shown to be associated with the development of gastric cancer and peptic ulcer diseases. Eradication of H. pylori infection reduces the risk of gastric cancer and the recurrence rate of peptic ulcer disease. However, the adverse effects, such as diarrhea and abdominal pain occurred in about 20-30% of patient during eradication therapies for H. pylori. Dysbiosis of the gut microbiota might contribute to the adverse effects.

Aims: Therefore, the investigators aimed to assess the efficacy of probiotic supplementation during the eradication therapy with 14-day sequential therapy in the reduction of adverse effects and the restoration of the dysbiosis.

Methods:

This will be a double-blind, placebo controlled, multi-center randomized trial. 200 patients with H. pylori infection naïve to eradication therapy will be enrolled.

Before First Line Treatment: Any two positive of CLO test, histology, serology and culture or a positive UBT will be considered as H. pylori infected.

After First Line Treatment: C13-UBT will be used to assess the existence of H. pylori 6-8 weeks after 14-day sequential therapy

Long term reinfection: C13-UBT will be used to assess the recurrence of H. pylori 1 year after14-day sequential therapy

Interventions: First line therapy: eligible patients will be randomized into one of the two groups.

Group (A): probiotic plus 14-day sequential therapy D1-D56: probiotics 1 pack bid for 56 days D1-D7: (esomeprazole + amoxicillin bid) for 7 days D8-D14: (esomeprazole + clarithromycin + metronidazole bid) for another 7 days

Group (B): placebo plus 14-day sequential therapy D1-D56: placebo 1 pack bid for 56 days D1-D7: (esomeprazole + amoxicillin bid) for 7 days D8-D14: (esomeprazole + clarithromycin + metronidazole bid) for another 7 days

Follow-up

1. The stool samples will be collected before, and 2 and 8 weeks and 1 year after eradication therapy to analyze the changes in the antibiotic resistance and microbiota of gut flora
2. The body weight, waist and hip circumference and serum lipid profile, sugar, and HBA1C levels will be collected before , and 2 and 8 weeks and 1 year after eradication therapy
3. Determination of antibiotic resistance of H. pylori: Agar dilution test will be used to determine the minimum inhibitory concentrations of antibiotics. Mutations in 23S rRNA will also be determined by PCR followed by direct sequencing

Outcome Measurement:

Primary End Point: Incidence of adverse effects in the first line therapy in the two treatment groups

Secondary End Point:

1. Eradication rates in the first line treatment in the two treatment groups
2. Changes of gut microbiota in the two treatment groups
3. Antibiotic resistance of gut flora after first line treatments in the two treatment groups
4. Re-infection rate one year after eradication therapy

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged greater than 20 years with H. pylori infection naïve to treatment are considered eligible for enrollment.

Exclusion Criteria:

* children and teenagers aged less than 20 years
* history of gastrectomy
* gastric malignancy, including adenocarcinoma and lymphoma
* previous allergic reaction to antibiotics (amoxicillin, metronidazole, clarithromycin, probiotics) and PPI (esomeprazole)
* contraindication to treatment drugs
* pregnant or lactating women
* severe concurrent disease
* concomitant use of clopidogrel
* unwilling to accept random assignment of subjects

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse effects in the first line therapy in the two treatment groups | 8 weeks
  At enrollment, the patients will be informed of the common side effects from the studied drugs and they will be asked to record these symptoms during treatment. A standardized interview and questionnaire will be used to assess the adverse events and compliance at the end of treatment. Patients with low compliance as defined by taking less than 80% of the pills and those lost to follow up will be excluded from the per-protocol analysis.

SECONDARY OUTCOMES:
Eradication rates in the first line treatment in the two treatment groups | 6 weeks
  Urea breath testing will be done at least 6 weeks after completion of eradication therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Jyh-Ming Liou, Taipei, Taiwan, Taiwan